CLINICAL TRIAL: NCT03353532
Title: Staphylococcus Aureus Surgical Site Infection Multinational Epidemiology in Europe
Acronym: SALT
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Oliver Cornely, MD, Prof. Dr., University of Cologne
Other Study IDs: SALT
Record Dates: First submitted 2017-11-20; First posted 2017-11-27 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Staphylococcus Aureus; Wound Infection, Surgical; Epidemiology
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort: Adult patients with SSI after any surgical procedure.
- Case-Control: Cases: Patients establishing S. aureus SSI Controls: Patients from the same center who did not undergo S. aureus SSI, matched by the following criteria
  * Type of procedure
  * Age
  * ASA score
  * BMI
  * Duration of procedure (as percentile for this procedure)
  * Diabetes
  * Sex

SUMMARY:
This is a retrospective multinational, multicenter cohort study with a nested case-control. The study includes all surgical procedures performed at a participating site to prevent bias.

Data will be assessed in two populations.

Cohort population: Export of electronic file data on demographics, surgical procedure ICPM code, duration of procedure, American Society of Anesthesiologists (ASA) score, body mass index, comorbidity ICD codes, and wound class of all patients undergoing surgery.

Nested case-control population: For patients establishing S. aureus SSI and 1:1 matched controls from the same center further data will be captured: Length of hospitalization, length of ICU stay and reason as well as attribution to SSI, survival at 30 and at 90 days, antibiotic treatments including duration, functional status at admission and at final discharge; necessity for surgical revision, and death attributed to SSI.

If readmission is necessary, reason and attribution to SSI, length of hospitalization and length of ICU stay as well as all antibiotic treatments and their duration will be recorded.

The cases causative pathogens including resistance patterns and type of SSI according to CDC criteria will be captured.

Matching criteria comprise the following:

* Type of procedure
* Age
* ASA score
* BMI
* Duration of procedure (as percentile for this procedure)
* Diabetes
* Sex

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of surgery

Exclusion Criteria:

* Cases with missing data defined as "missing completely at random" (MCAR)
* Infection at the time of surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with SSI after any surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 178902 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
To determine overall incidence of Staphylococcus aureus surgical site infections in Europe | 30 days from surgical procedure
  Surgical site infections will be determined within the cohort of all patients that underwent surgery within 1 year at all participating sites.
To determine procedure specific incidence of Staphylococcus aureus surgical site infections in Europe | 30 days from surgical procedure
  Surgical site infections will be determined within the cohort of all patients that underwent surgery within 1 year at all participating sites. A subgroup Analysis will reveal procedure specific incidence.

SECONDARY OUTCOMES:
To determine the overall outcomes of Staphylococcus aureus surgical site infections in Europe | 30 days from surgical procedure
  The Outcome will be assessed within the case-control part and achieved by comparison of Overall Outcome of cases and controls
To determine the procedure specific outcomes of Staphylococcus aureus surgical site infections in Europe | 30 days from surgical procedure
  The Outcome will be assessed within the case-control part and achieved by comparison of procedure specific Outcome of cases and controls
To determine the overall economic burden of Staphylococcus aureus surgical site infections in Europe | 30 days from surgical procedure
  The economic burden will be assessed within the case-control part and achieved by comparison of Overall economic burden (i.e. ICU Treatment, hemodialysis and mechanical Ventilation) of cases and controls
To determine the procedure specific economic burden of Staphylococcus aureus surgical site infections in Europe | 30 days from surgical procedure
  The economic burden will be assessed within the case-control part and achieved by comparison of procedure specific economic burden (i.e. ICU Treatment, hemodialysis and mechanical Ventilation) of cases and controls

OTHER OUTCOMES:
To characterize the composition of the surgical patient population in Europe | 30 days from surgical procedure
  The composition of the surgical patient population in Europe will be performed by subgroup Analysis of the cohort
To estimate the number of patients at risk for Staphylococcus aureus surgical site infection | 30 days from surgical procedure
  This will be extrapolated from epidemiologcal data assessed within the cohort
To estimate the economic burden, including direct treatment and indirect costs, imposed by Staphylococcus aureus surgical site infections in Europe | 30 days from surgical procedure
  Direct and indirect Treatment costs will be assessed within the case-control part. Cases and controls will be compared regarding costs.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A Cornely, MD, Principal Investigator — University of Cologne
Locations (14):
- France (3):
  - Centre Hospitalier Départemental Vendee, La Roche-sur-Yon
  - Centre Hospitalier et Universitaire de Limoges, Limoges
  - Centre Hospitalier Régional et Universitaire de Tours, Tours
- Germany (4):
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - University Hospital Bonn, Bonn
  - Jena University Hospital, Jena
  - Hospital of the University of Munich, Munich
- University of Udine and Azienda Sanitaria Universitaria Integrata, Udine, Italy
- Spain (5):
  - Hospital Clínic Barcelona, Barcelona
  - Institut Hospital del Mar d'Investigacions Mèdiques, Barcelona
  - Hospital General Universitario Gregorio Marañón e Instituto de Investigación Sanitaria Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia
- Manchester University NHS Foundation Trust (MFT), Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mellinghoff SC, Bruns C, Albertsmeier M, Ankert J, Bernard L, Budin S, Bataille C, Classen AY, Cornely FB, Couve-Deacon E, Fernandez Ferrer M, Fortun J, Galar A, Grill E, Guimard T, Hampl JA, Wingen-Heimann S, Horcajada JP, Kohler F, Koll C, Mollar J, Munoz P, Pletz MW, Rutz J, Salmanton-Garcia J, Seifert H, Serracino-Inglott F, Soriano A, Stemler J, Vehreschild JJ, Vilz TO, Naendrup JH, Cornely OA, Liss BJ. Staphylococcus aureus surgical site infection rates in 5 European countries. Antimicrob Resist Infect Control. 2023 Sep 19;12(1):104. doi: 10.1186/s13756-023-01309-w. PMID 37726843
- [Derived] Mellinghoff SC, Bruns C, Al-Monajjed R, Cornely FB, Grosheva M, Hampl JA, Jakob C, Koehler FC, Lechmann M, Maged B, Otto-Lambertz C, Rongisch R, Rutz J, Salmanton-Garcia J, Schlachtenberger G, Stemler J, Vehreschild J, Wulfing S, Cornely OA, Liss BJ. Harmonized procedure coding system for surgical procedures and analysis of surgical site infections (SSI) of five European countries. BMC Med Res Methodol. 2022 Aug 12;22(1):225. doi: 10.1186/s12874-022-01702-w. PMID 35962320
- [Derived] Mellinghoff SC, Vehreschild JJ, Liss BJ, Cornely OA. Epidemiology of Surgical Site Infections With Staphylococcus aureus in Europe: Protocol for a Retrospective, Multicenter Study. JMIR Res Protoc. 2018 Mar 12;7(3):e63. doi: 10.2196/resprot.8177. PMID 29530837